CLINICAL TRIAL: NCT00073073
Title: A Trial of Exemestane in Postmenopausal Women With DCIS or at High Risk for Invasive Breast Cancer
Brief Title: Exemestane and Celecoxib in Postmenopausal Women at High Risk for Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 040044; 04-C-0044 (Other: NCI); NCT00085072 (obsolete NCT alias)
Record Dates: First submitted 2003-11-14; First posted 2003-11-17 (Estimated); Results first posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2015-10

CONDITIONS: Breast Neoplasms
Keywords: Chemoprevention; Mammographic Density; Bone Mineral Density; Biomarkers; Safety; Breast Cancer; Postmenopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Calcium Carbonate; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exemestane (Experimental): exemestane 25 mg by mouth (PO) every day for two years taken with calcium carbonate 1200 mg PO every day and vitamin D 400 IU PO every day Initially patients were initially planned to receive Celecoxib but the study was amended prior to any subject going on and Celecoxib was never administered to any subjects.
  Interventions: Drug: Exemestane; Dietary Supplement: Calcium carbonate; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Exemestane — exemestane 25 mg by mouth (PO) every day for two years
  Other Names: Aromasin
Dietary Supplement: Calcium carbonate — calcium carbonate 1200 mg PO every day x 2 years
Dietary Supplement: Vitamin D — Vitamin D 400 international units PO every day x 2 years

SUMMARY:
The primary goal of this 5-year study is to determine whether exemestane alone or in combination with celecoxib decreases breast tissue density in healthy postmenopausal women at high risk for breast cancer. Dense breast tissue seen on mammography has been linked to an increased risk of breast cancer. The study will also examine the effects of exemestane and celecoxib on bone density, blood hormone levels and quality of life. Exemestane, approved by the Food and Drug Administration for treating postmenopausal women with breast cancer, lowers the amount of estrogen in the body. Celecoxib, approved for treating arthritis pain and for reducing the number or colon polyps in an inherited syndrome, is an anti-inflammatory drug. Half of the women in the study will receive exemestane alone and half will receive exemestane and celecoxib together.

In December 2004, the arm using exemestane and celecoxib was closed to accrual

Postmenopausal women who are at increased risk for developing invasive breast cancer may be eligible to participate. Candidates are screened with breast cancer risk assessment, medical history and physical examination, blood tests, review of medical records, if needed, breast biopsy, and dual energy x-ray absorptiometry (DEXA) scan to assess bone density. For the DEXA scan, the subject lies still on a table for about 30 minutes while the spine and hip are scanned using a small amount of radiation.

Participants take exemestane in pill form once a day for 2 years. They also take calcium and vitamin D pills daily to help protect bone health. They are followed in the clinic during the course of the study to determine the amount of drug taken and any side effects, and for the following tests and procedures:

* Medical evaluation and blood tests at after 1 and 3 months on study drugs
* Medical evaluation at 6 months
* Breast biopsy at screening and then at 12 months
* dual-emission x-ray absorptiometry (DEXA) scan of the spine, mammogram and routine blood tests before starting study drugs and then yearly for 5 years.

DETAILED DESCRIPTION:
Background:

Evidence from adjuvant treatment trials of invasive breast cancer with aromatase inhibitors suggests that these agents are superior to tamoxifen in preventing contralateral breast cancer and are well tolerated. These agents are promising breast cancer chemopreventive agents. Data on safety and effect on surrogate biomarkers in a healthy at risk population is lacking.

Objectives:

Primary:

-The primary objective is to evaluate the study drug effects on mammographic density after one year on treatment.

Secondary:

-Secondary objectives include assessing the effect of the intervention on bone mineral density, serum hormones and lipids, and breast tissue biomarkers.

Eligibility:

Eligible patients are postmenopausal women who meet one of the following criteria:

* History of stage I or II breast cancer 2 years out from definitive therapy.
* Gail model 5 year risk greater than or equal to 1.7%
* History of treated ductal carcinoma in-situ (DCIS)
* History of high risk lesion on breast biopsy (atypical ductal hyperplasia (ADH), atypical lobular hyperplasia (ALH), lobular carcinoma in-situ (LCIS))
* Known or suspected breast cancer 1, early onset (BRCA1) or breasts cancer 2, early onset (BRCA2) mutation
* Subjects must have adequate bone mineral density by dual-emission x-ray absorptiometry (DEXA) scan in order to enroll.

Design:

* This is an open label study of exemestane in postmenopausal women with an elevated risk of developing invasive breast cancer. Forty five subjects will be enrolled and receive standard dose exemestane (25 mg each day (QD)), calcium and vitamin D.
* Each subject will continue treatment for a total of two years.
* Changes in mammographic breast density and bone mineral density will be evaluated annually which will provide long term biomarker and safety information about prevention therapy with exemestane.

ELIGIBILITY:
* INCLUSION CRITERIA:

Postmenopausal female.

Postmenopausal defined as no menses for at least 12 months or bilateral oophorectomy. In unclear cases, (e.g. 50 year old who has had hysterectomy) chemical confirmation of postmenopausal status may be confirmed with follicle stimulating hormone (FSH) greater than 35 U/L.

Elevated risk for developing invasive breast cancer by virtue of one of the following criteria:

Gail Model risk of greater than or equal to 1.7% over 5 years from study entry. (This is the same minimum level of risk required for a subject to be eligible for the recently completed NSABP-P1 tamoxifen breast cancer prevention trial).

Lobular neoplasia.

Atypical ductal hyperplasia.

DCIS (ductal carcinoma in situ) that has been previously treated with mastectomy or lumpectomy and radiation, +/- tamoxifen.

Deleterious mutations in BRCA1 or 2 OR A priori risk assessment of 20% chance or greater of carrying BRCA1/2 gene mutation. The BRCAPRO and Couch model will both be used to asses this risk. If a woman has a 20% risk of carrying a BRCA1/2 mutation by either model, she will meet eligibility criteria.

Prior stage I or II breast cancer at least 2 years out from treatment for invasive disease and no prior use of aromatase inhibitors.

Subjects should be willing to abstain from use of hormonal therapies (e.g. tamoxifen, hormone replacement therapy, oral contraceptive pills, hormone-containing intrauterine devices (IUDs). E-string is acceptable). Venlafaxine will be offered as supportive care for women with menopausal symptoms.

Eastern Cooperative Oncology Group (ECOG) performance status 0-1.

Subject has been counseled regarding her options and has signed the informed consent document.

Baseline dual-emission x-ray absorptiometry (DEXA) scan with bone mineral density (BMD) T-score greater than or equal to 2.5 at antero posterior (AP) spine.

Hemoglobin greater than or equal to 11 g/dl.

Creatinine less than 1.5 times the upper limits of normal.

Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) less than 2.5 times upper limit of normal.

No investigational agent for the past 30 days.

If history of cancer (other than squamous or basal cell skin cancers), subject must have no evidence of disease at time of enrollment AND no history of cancer directed treatment in the 2 years preceding enrollment.

EXCLUSION CRITERIA:

Current or recent chronic use (within 3 months) of hormonal medications, e.g. oral contraceptive pills, hormone replacement therapy, tamoxifen, raloxifene, IUD with progestins or corticosteroids. (Subjects on chronic topical or inhaled steroids will be eligible for the study.) Current use of phenytoin, carbamazepine, rifampin due to increased estrogen metabolism.

History of clotting or bleeding disorder.

History of allergic reactions attributed to compounds of similar chemical or biologic composition to exemestane (e.g. anastrozole, letrozole, formestane).

Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suparna B Wedam, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (2):
- United States (2):
  - Lombardi Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Fisher B, Costantino JP, Wickerham DL, Redmond CK, Kavanah M, Cronin WM, Vogel V, Robidoux A, Dimitrov N, Atkins J, Daly M, Wieand S, Tan-Chiu E, Ford L, Wolmark N. Tamoxifen for prevention of breast cancer: report of the National Surgical Adjuvant Breast and Bowel Project P-1 Study. J Natl Cancer Inst. 1998 Sep 16;90(18):1371-88. doi: 10.1093/jnci/90.18.1371. PMID 9747868
- [Background] Baum M, Budzar AU, Cuzick J, Forbes J, Houghton JH, Klijn JG, Sahmoud T; ATAC Trialists' Group. Anastrozole alone or in combination with tamoxifen versus tamoxifen alone for adjuvant treatment of postmenopausal women with early breast cancer: first results of the ATAC randomised trial. Lancet. 2002 Jun 22;359(9324):2131-9. doi: 10.1016/s0140-6736(02)09088-8. PMID 12090977
- [Background] Jones S, Vogel C, Arkhipov A, Fehrenbacher L, Eisenberg P, Cooper B, Honig S, Polli A, Whaley F, di Salle E, Tiffany J, Consonni A, Miller L. Multicenter, phase II trial of exemestane as third-line hormonal therapy of postmenopausal women with metastatic breast cancer. Aromasin Study Group. J Clin Oncol. 1999 Nov;17(11):3418-25. doi: 10.1200/JCO.1999.17.11.3418. PMID 10550136
- [Derived] Gatti-Mays ME, Venzon D, Galbo CE, Singer A, Reynolds J, Makariou E, Kallakury B, Heckman-Stoddard BM, Korde L, Isaacs C, Warren R, Gallagher A, Eng-Wong J. Exemestane Use in Postmenopausal Women at High Risk for Invasive Breast Cancer: Evaluating Biomarkers of Efficacy and Safety. Cancer Prev Res (Phila). 2016 Mar;9(3):225-33. doi: 10.1158/1940-6207.CAPR-15-0269. Epub 2016 Jan 12. PMID 26758879
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-C-0044.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exemestane
Started | 46
Completed | 42
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Patients who were treated
Arm/Group | Exemestane
Number analyzed (Participants) | 42
Age, Continuous [Mean (Full Range); unit: years] | 59.1 [45 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Mammographic Density at 1 Year on Exemestane
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Exemestane
Number analyzed (Participants) | 42
percent change from baseline | -2.4 [-5.0 to 0.1]

2. Secondary Outcome: Effect of This Drug on Bone Mineral Density
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Exemestane
Number analyzed (Participants) | 42
percent change from baseline | -1.4 [-2.5 to -0.3]

3. Secondary Outcome: Change in Breast Density at 2 Years
Time Frame: 2 years
Measure: Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Exemestane
Number analyzed (Participants) | 42
percent change from baseline | -4.1 [-7.2 to -1.1]

4. Secondary Outcome: Effect of This Drug on Serum Hormones, Insulin-like Growth Factor Pathway Components, and Leptin at 3 Months and 1 Year
Time Frame: 3 months and 1 year
Population: Data were not collected
Arm/Group | Exemestane
Number analyzed (Participants) | 0

5. Secondary Outcome: Absolute Change of Lipid Profiles on Exemestane From Baseline
Time Frame: 1 year
Population: Change in total cholesterol
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Exemestane
Number analyzed (Participants) | 42
mg/dl | 181.6 (35.9)

6. Secondary Outcome: Effect of This Drug on Breast Tissue Trefoil Factor 1 and Proliferating Cell Nuclear Antigen Expression, Prolactin, and Breast Tissue Prolactin Receptor at 1 Year
Time Frame: 1 year
Population: Change in breast tissue trefoil factor 1
Measure: Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Exemestane
Number analyzed (Participants) | 35
percent change from baseline | -1.32 [-1.87 to -0.76]

7. Secondary Outcome: Effect of Exemestane on Autocrine Prolactin and Breast Tissue Prolactin Receptor at One Year
Time Frame: 1 year
Population: Outcome not measured
Arm/Group | Exemestane
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Serum and Breast Tissue Samples Collected for Exploratory Proteomic Profiles at One Year
Time Frame: 1 year
Population: Outcome not measured
Arm/Group | Exemestane
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Exemestane
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 41/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=42)
Hot flashes (Endocrine disorders) | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Vaginal dryness (Reproductive system and breast disorders) | 4
Fatigue (General disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Diarrhea (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No